CLINICAL TRIAL: NCT00166452
Title: Multicenter, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Lenalidamide in the Treatment of Complex Regional Pain Syndrome Type1
Brief Title: A Study of the Effect of Lenalidamide on Complex Regional Pain Syndrome Type 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Elgene Chemical (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 422-05
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Complex Regional Pain Syndrome, Type 1
MeSH Terms: conditions — Complex Regional Pain Syndromes

INTERVENTIONS:
Drug: Lenalidamide

SUMMARY:
The purpose of this study is to determine if lenalidomide is a safe and effective treatment for complex regional pain syndrome type 1 (CRPS).

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = to 18 years
2. Signed consent form
3. A diagnosis of CRPS type I for at least one-year duration with unilateral involvement of a distal limb
4. CRPS pain intensity score at least 4 on an 11-point PI-NRS
5. Measurable sural, median sensory, median motor and peroneal motor nerve conductions
6. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days of starting the study drug. They must agree to use adequate contraceptive methods not including steroid-based contraceptives. They must also agree to have pregnancy tests every 4 weeks while on the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-07; Primary Completion 2007-04 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
RPS Pain Intensity Numeric Rating Scale (PI-NRS): At least 30% reduction from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Keith A Bengtson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States